CLINICAL TRIAL: NCT01584492
Title: Double Blind, Double Dummy, Cross-over Study to Compare the Bronchodilator Effect of CHF1535 pMDI (Fixed Combination of Beclometasone 50 µg + Formoterol 6 µg) Versus Free Combination of Beclometasone Plus Formoterol pMDI in Asthmatic Children
Brief Title: Bronchodilator Effect of CHF1535 pMDI Versus Free Combination of Beclometasone Plus Formoterol pMDI in Asthmatic Children
Acronym: PAED3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-0903-PR-0060; 2011-002060-24 (EudraCT Number)
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Beclomethasone; Albuterol; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Treatment A (Experimental): CHF 1535 50/6 administered via a pMDI with spacer, 1 inhalation (dose: BDP 50 µg/FF 6 µg) + placebo HFA pMDI with spacer, 5 inhalations in the morning at the clinic
  Interventions: Drug: beclomethasone+formoterol 50/6 (1 inhalation)
- Treatment B: (Experimental): CHF 1535 50/6 administered via a pMDI with spacer, 2 inhalations (dose: BDP 100 µg/FF 12 µg) + placebo HFA pMDI with spacer, 4 inhalations in the morning at the clinic
  Interventions: Drug: CHF 1535 50/6 (2 inhalations)
- Treatment C (Experimental): CHF 1535 50/6 (dose: BDP 200 µg/FF 24 µg) administered via a pMDI with spacer, 4 inhalations (dose: BDP 200 µg/FF 24 µg) in the morning at the clinic + placebo HFA pMDI with spacer, 2 inhalations in the morning at the clinic
  Interventions: Drug: CHF 1535 50/6 (4 inhalations)
- Treatment D (Active Comparator): formoterol 6 µg HFA administered via a pMDI with spacer, 2 inhalations (dose: FF 12 µg) + extrafine BDP 50 µg, administered via a pMDI with spacer, 2 inhalations (dose: BDP 100 µg), in the morning at the clinic + placebo HFA pMDI with spacer, 2 inhalations in the morning at the clinic
  Interventions: Drug: Formoterol + Beclomethasone dipropionate
- Treatment E (Placebo Comparator): placebo pMDI with spacer, 6 inhalations in the morning at the clinic
  Interventions: Drug: Placebo (6 inhalations)

INTERVENTIONS:
Drug: beclomethasone+formoterol 50/6 (1 inhalation) — CHF 1535 50/6 (fixed combination of extrafine beclomethasone dipropionate 50 µg + formoterol fumarate 6 µg/metered dose) administered via a pMDI with spacer
  Other Names: CHF1535, Atimos®, Ventolair®, Ventolin®
  Arms: Treatment A
Drug: CHF 1535 50/6 (2 inhalations) — CHF 1535 50/6 (fixed combination of extrafine beclomethasone dipropionate 50 µg + formoterol fumarate 6 µg/metered dose) administered via a pMDI with spacer
  Other Names: CHF1535, Atimos®, Ventolair®, Ventolin®
  Arms: Treatment B:
Drug: CHF 1535 50/6 (4 inhalations) — CHF 1535 50/6 (fixed combination of extrafine beclomethasone dipropionate 50 µg + formoterol fumarate 6 µg/metered dose) administered via a pMDI with spacer
  Other Names: CHF1535, Atimos®, Ventolair®, Ventolin®
  Arms: Treatment C
Drug: Formoterol + Beclomethasone dipropionate — * Formoterol HFA pMDI 6 µg / actuation
  * Extrafine BDP HFA pMDI 50 µg/actuation
  Other Names: CHF1535, Atimos®, Ventolair®, Ventolin®
  Arms: Treatment D
Drug: Placebo (6 inhalations) — Matched placebo via pMDI
  Other Names: CHF1535, Atimos®, Ventolair®, Ventolin®
  Arms: Treatment E

SUMMARY:
The purpose of this clinical study is to compare the improvement in breathing of single administration of CHF 1535 50/6 pMDI (fixed combination of a corticosteroid drug beclomethasone 50 µg + formoterol 6 µg/puff, 2 inhalations, total dose 100/12 µg) given with spacer versus free combination of beclomethasone 50 µg/puff pMDI (2 inhalations, total dose 100 µg) given with spacer plus formoterol 6 µg/puff pMDI (2 inhalations, total dose 12 µg) given with spacer in terms of FEV1 from 0 to 12 hours in asthmatic children.

Additionally the study aims to evaluate the effects of doses of CHF 1535 pMDI compared to placebo and the effect on other lung function parameters, to assess the safety and tolerability of CHF 1535 dosages in children.

DETAILED DESCRIPTION:
FEV1 from 0 to 12 hours standardised by time will be statistically analysed taking into account treatment, period and subject and pre-dose FEV1.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the parents/legal representatives and/or the subject (if and when appropriate)
* Prepuberal male and female outpatients, aged ≥ 5 and < 12 years (Tanner stage I and II)
* Clinical diagnosis of asthma according to Global Strategy for Asthma Management and Prevention (GINA) revised version 2009 at least six months prior to screening visit.
* Already treated with inhaled short acting Beta2-agonists as required and / or inhaled beclomethasone dipropionate up to 400 µg or equivalent.
* Forced Expiratory Volume during the first second (FEV1) ≥ 60% and ≤ 95% of predicted normal values at the screening visit.
* A documented positive response to the reversibility test at the screening visit, defined as Delta FEV1 ≥ 15% over baseline, 15 minutes after 400 μg salbutamol pressurised Meter Dose Inhaler (ATS/ERS taskforce 2005).
* A cooperative attitude and ability to use a pMDI and a spacer (Aerochamber Plus and Volumatic).

Exclusion Criteria:

* Endocrinological diseases or other chronic diseases.
* Known sensitivity to the components of study medication.
* Any concomitant disease requiring additional treatment with topic or systemic glucocorticosteroids.
* Allergy to one component of medications used.
* Intolerance or contra-indication to treatment with Beta2-agonists and/or inhaled corticosteroids.
* Having received an investigational drug within 2 months before the current study.
* Inability to comply to study procedures or to study treatment intake.
* Occurrence of acute asthma exacerbations or respiratory tract infections in the 4 weeks preceding the screening visit.
* Significant seasonal variation in asthma or asthma occurring only during episodic exposure to an allergen or a chemical sensitizer.
* History of cystic fibrosis, bronchiectasis or alpha-1 antitrypsin deficiency.
* History of near fatal asthma (e.g. brittle asthma, hospitalisation for asthma exacerbation in Intensive Care Unit).
* Diagnosis of restrictive lung disease.
* Significant medical history and/or treatments for cardiac, renal, neurological, hepatic, endocrine diseases, or any laboratory abnormality indicative of a significant underlying condition, that may interfere with patient's safety, compliance, or study evaluations, according to the investigator's opinion.
* QTc interval (Fridericia's formula) higher than 450 msec at screening visit

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2011-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
bronchodilator effect of test treatment | FEV1 AUC measured over 12 hours
  To compare the bronchodilator effect of single administration of CHF 1535 50/6 pMDI (fixed combination of extrafine beclomethasone dipropionate 50 µg + formoterol fumarate 6 µg/metered dose, 2 inhalations, total dose 100/12 µg) given with spacer vs. free combination of extrafine beclomethasone dipropionate 50 µg/metered dose pMDI (2 inhalations, total dose 100 µg) given with spacer plus formoterol 6 µg/metered dose pMDI (2 inhalations, total dose 12 µg) given with spacer in terms of FEV1 AUC 0-12 hours corrected by time for the 12 hours study period in asthmatic children.

SECONDARY OUTCOMES:
dose-related effects of test treatment | Peak FEV1 and FEV1 measured at 12 hours post-dose
  To evaluate the dose-related effects of CHF 1535 pMDI compared to placebo and the effect on other lung function parameters, to assess the safety and tolerability of CHF 1535 regimens in children.

CONTACTS AND LOCATIONS:
Overall Officials: Petr Pohunek, M.D., Principal Investigator — Charles University, 2nd Medical Faculty and University Hospital Motol - CZECH REPUBLIC
Locations (2):
- Poradnia Alergologiczna, Dębica, Debica, Poland, Poland
- Zaporizhzhia State Medical University, Zaporizhzhia, Zaporizhzhia Oblast, Ukraine

REFERENCES:
- [Derived] Pohunek P, Varoli G, Reznichenko Y, Mokia-Serbina S, Brzostek J, Kostromina V, Kaladze M, Muraro A, Carzana E, Armani S, Kaczmarek J. Bronchodilating effects of a new beclometasone dipropionate plus formoterol fumarate formulation via pressurized metered-dose inhaler in asthmatic children: a double-blind, randomized, cross-over clinical study. Eur J Pediatr. 2021 May;180(5):1467-1475. doi: 10.1007/s00431-020-03888-x. Epub 2021 Jan 6. PMID 33404895
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2011-002060-24